CLINICAL TRIAL: NCT06676098
Title: The Optimal Injection Site for a 3D Guided Inferior Alveolar Nerve Block Device (IANBD): A Randomized Control Trial
Brief Title: The Optimal Injection Site for a 3D Guided Inferior Alveolar Nerve Block Device (IANBD)
Acronym: IANBD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-43160
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Inferior Alveolar Nerve Block
Keywords: Inferior alveolar nerve block (IANB); Inferior alveolar nerve block device (IANBD); 3D guided IANBD; Cone beam computed tomography (CBCT)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IANBD guided Inferior Alveolar Nerve block (IANB) injection (Experimental): Participants will receive a guided IANB using an IANBD.
  Interventions: Procedure: IANBD 3D guided approach

INTERVENTIONS:
Procedure: IANBD 3D guided approach — The IANBD will be used to administer the dental anesthetic 2mm medial to the lingula

SUMMARY:
Given the thicker cortical bone in the mandible compared to the maxilla, mandibular teeth cannot be effectively anesthetized via local infiltration anesthesia. Instead, clinicians typically perform regional anesthesia and most commonly, Inferior Alveolar Nerve block (IANB). However, the inferior alveolar nerve is deeply submerged by surrounding structures of bone, muscles, ligaments and vessels. Traditional IANB is a technique by using anatomical landmarks not directly related to Inferior Alveolar Nerve (IAN) to approximate the location of mandibular foramen, where IAN enters mandible. IANB is considered a blind technique and known for the lack of accuracy and precision. The failure rate can be as high as 30-45%. In contrast, the investigator's cone beam computed tomography (CBCT) guided IANB device (IANBD) effectively directs the needle to the mandibular foramen which improves the success rate of the IANB on the first attempt, minimizes injection tissue damage, and reduces patient discomfort.

In this proof of concept trial, a 3D printed CBCT guided IANBD will be used to administer anesthesia at three injection sites instead of the traditional IANB technique. Participants will be consented patients at the postdoctoral endodontic treatment center, Department of Endodontics, Boston University (BU) Henry M. Goldman School of Dentistry.

The goal of this research is to to evaluate the acceptability, safety, and effectiveness of guided anesthesia using the IANBD by enrolling 10 subjects who require non-surgical endodontic therapy with a simple, affordable and reliable prototype to be used by clinicians in the dental care setting.

ELIGIBILITY:
Inclusion Criteria:

* Patient of Henry M. Goldman School of Dentistry (GSDM)
* Medical History indicating American Society of Anesthesiology (ASA)1
* Need Non-surgical Endodontic Therapy on Mandibular Molar or Premolar
* Asymptomatic pulpal diagnosis (normal, necrotic, asymptomatic irreversible pulpitis, retreatment with no symptoms)
* The quadrant to be treated must have at least 3 vital teeth.
* Going to receive a CBCT required for clinical purposes
* Must be willing to receive guided IANB

Exclusion Criteria:

* Allergy to lidocaine or articaine
* Resin allergy
* Normal teeth unresponsive to thermal testing (ie calcified chamber)
* Prior jaw surgery
* Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Participant acceptability | 30 minutes post dental procedure
  For this proof of concept trial, the investigators developed a questionnaire with 3 open-ended questions asking participants; 1) did they have mandibular anesthesia before for a dental procedure and if yes how did this compare, 2) was the size of the device acceptable, and 3) was the taste of the device acceptable. The responses will be assessed to determine if overall the IANBD was acceptable or not to each participant.
Clinician acceptability | 30 minutes post dental procedure
  For this proof of concept trial, the investigators developed a questionnaire with 5 open-ended questions asking clinicians; 1) how easy was it to set up the IANBD, 2) how time consuming was it to use the IANBD, 3) could you visualize the needle with the device, 4) are you likely to switch to the IANBD, and 5) compare this technique with previous IANB methods. The responses will be assessed to determine if overall the IANBD was acceptable or not to each clinician.
Safety of IANBD based on number of adverse events | at the end of the study, about 2 years
  The number of adverse events that occur will be abstracted from records of the procedure for each participant.
Safety of IANBD based on type of adverse events | at the end of the study, about 2 years
  The types of adverse events that occur will be abstracted from records of the procedure for each participant.

SECONDARY OUTCOMES:
Pulp vitality | baseline, 1 minute, 4 minutes, 7 minutes, 10 minutes, 13 minutes
  The Cold test will be done to assess pulpal vitality/anesthesia. If the Cold test is negative, the anesthesia is successful.

CONTACTS AND LOCATIONS:
Overall Officials: Tum-Yi Hsu, DMD DScD, Principal Investigator — BU Goldman School of Dental Medicine, Endodontics
Locations (1):
- Goldman School of Dental Medicine, Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No